CLINICAL TRIAL: NCT04094870
Title: Z 31801 - A Pilot Trial of Perinatal Depression Treatment in HIV Infected Women
Brief Title: A Pilot Trial of Perinatal Depression Treatment in HIV Infected Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-3411; 1R21MH115806 (NIH); Z 31801 (Other: UNC)
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2020-12

CONDITIONS: Perinatal Depression; HIV-1-infection
Keywords: perinatal depression; HIV; Antiretroviral Treatment; Interpersonal psychotherapy
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Intervention Model Description: Daily self-administered selective serotonin reuptake inhibitor (SSRI) Sertraline initial dose of 25 mg tablet versus IPT in a 1:1 ratio commenced between six and 8 weeks postpartum and continued through 30 weeks postpartum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Antidepressant medication (Active Comparator): Daily self-administered selective serotonin reuptake inhibitor (SSRI) Sertraline 25 mg table
  Interventions: Drug: Sertraline
- Interpersonal therapy (Active Comparator): Up to 11 planned therapy sessions over a 24-week period beginning the day of randomization
  Interventions: Behavioral: Interpersonal therapy

INTERVENTIONS:
Drug: Sertraline — daily SSRI (Sertraline 25mg)
  Other Names: SSRI
  Arms: Antidepressant medication
Behavioral: Interpersonal therapy — 11 sessions over a 24-week period
  Arms: Interpersonal therapy

SUMMARY:
This pilot study will evaluate, through quantitative and qualitative methods, whether different treatments for postpartum depression are feasible and acceptable in postpartum HIV infected women on antiretrovirals (ART). The study will take place at several clinics in Lusaka, Zambia.

DETAILED DESCRIPTION:
The standard of care for treating postpartum depression in the US is antidepressants, psychotherapy or both. Little data exist on the best method for treating perinatal depression (PND) in Sub-Saharan Africa. This is a mixed method study including a pilot randomized controlled trial (RCT) of antidepressant medication (ADM) versus interpersonal psychotherapy (IPT) and qualitative semi-structured interviews (SSIs). The study will enroll 100 pregnant HIV infected women over the age of 18 seeking postnatal care and continuing antiretroviral therapy in pregnancy. An additional 20 women enrolled in the RCT will be invited to participate in SSIs. Each participant will be followed for 24 weeks.

ELIGIBILITY:
Inclusion criteria:

* 18 years of age or older
* Documentation of confirmed HIV-1 infection
* Six to eight weeks postpartum
* Currently taking ART treatment
* Able and willing to provide written informed consent
* Willing to adhere to study visit schedule
* PND diagnosis confirmed by Mini-International Neuropsychiatric Interview

Exclusion criteria:

* Taking an ADM in the prior 12 months prior to enrollment
* Actively suicidal
* Known or suspected allergy or contraindication to first line Sertraline
* Any other condition (social or medical) which, in the opinion of the study staff, would make trial participation unsafe or complicate data interpretation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stringer, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- Zambia (2):
  - Kamwala District Health Centre, Lusaka
  - University Teaching Hospital, Lusaka

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: Investigator who proposes to use the data has IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Spelke MB, Paul R, Blette BS, Meltzer-Brody S, Schiller CE, Ncheka JM, Kasaro MP, Price JT, Stringer JSA, Stringer EM. Interpersonal therapy versus antidepressant medication for treatment of postpartum depression and anxiety among women with HIV in Zambia: a randomized feasibility trial. J Int AIDS Soc. 2022 Jul;25(7):e25959. doi: 10.1002/jia2.25959. PMID 35803896

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Antidepressant Medication | Interpersonal Therapy
Started | 40 | 40
Completed | 39 | 39
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antidepressant Medication | Interpersonal Therapy | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (5.5) | 30.0 (5.3) | 29.7 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 40 | 40 | 80
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 40 | 40 | 80
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Zambia | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Women Approached Who Agreed to Pre-Screening With EPDS
Description: In order to determine feasibility, the number of women who agree to be pre-screened with the Edinburgh Postnatal Depression Screen (EPDS) within 2-7 weeks postpartum
Time Frame: 2-7 weeks postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Approached Patients: Eligible patients approached for participation
Arm/Group | Approached Patients
Number analyzed (Participants) | 240
Participants | 240

2. Primary Outcome: Number of Women Pre-Screened Who Have an EPDS Score >/= 6
Description: The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report used to measure postpartum depression with score range 0-30, a higher score indicates greater symptom burden. A score of >/= 6 is indicative of a woman being at risk of perinatal depression. The number of women with an EPDS >/= 6 out of all of the women who were pre-screened with an EPDS.
Time Frame: 2-7 weeks postpartum
Measure: Count of Participants; unit: Participants
Groups:
- Approached Patients Who Completed Pre-Screening EPDS: Potentially eligible patients who underwent pre-screening with EPDS
Arm/Group | Approached Patients Who Completed Pre-Screening EPDS
Number analyzed (Participants) | 240
Participants | 199

3. Primary Outcome: Number of Women With an EPDS >/= to 6 Who Were Consented and Underwent Diagnostic Testing With MINI
Description: MINI International Neuropsychiatric Interview (MINI) is a brief structured diagnostic interview and is designed to assess the most common psychiatric disorders in ICD-10 and DSM-5. MINI modules were used: major depressive disorder and generalized anxiety disorder. Questions are rated dichotomously (yes/no) and clinical judgment should be used in coding the responses, asking for examples if needed. Participants will be eligible for the study if they are diagnosed with depression or anxiety based on the MINI assessment. After pre screening with an EPDS, women with an EPDS >/=6 were invited to undergo MINI diagnostic testing after signed consent.
Time Frame: 2-7 weeks postpartum
Population: 199 women were eligible for the MINI based on an EPDS >/= 6.
Measure: Count of Participants; unit: Participants
Groups:
- All Participants With an EPDS >/=6: Women eligible for the MINI based on an EPDS >/=6
Arm/Group | All Participants With an EPDS >/=6
Number analyzed (Participants) | 199
Participants | 120

4. Primary Outcome: Number of Women With Anxiety or Depression Based on the MINI Who Agree to Participate in the Study
Description: MINI International Neuropsychiatric Interview (MINI) is a brief structured diagnostic interview and is designed to assess the most common psychiatric disorders in ICD-10 and DSM-5. MINI modules were used: major depressive disorder and generalized anxiety disorder. Questions are rated dichotomously (yes/no) and clinical judgment should be used in coding the responses, asking for examples if needed. Participants will be eligible for the study if they are diagnosed with depression or anxiety based on the MINI assessment.
Time Frame: 6-8 weeks postpartum
Population: 91 met diagnostic criteria by MINI.
Measure: Count of Participants; unit: Participants
Groups:
- Women Who Met Diagnostic Criteria by MINI and Agreed to Participate in the Study: Eligible women diagnosed with anxiety or depression based on the MINI who agree to participate
Arm/Group | Women Who Met Diagnostic Criteria by MINI and Agreed to Participate in the Study
Number analyzed (Participants) | 91
Participants | 80

5. Primary Outcome: Number of Women Retained in the Study
Description: Number of women who are enrolled in the study who complete the final study visit
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antidepressant Medication | Interpersonal Therapy
Number analyzed (Participants) | 40 | 40
Participants | 39 | 39

6. Secondary Outcome: Number of Women With an EPDS Score Decline of 3 Points From Baseline
Description: The Edinburgh Postnatal Depression Scale (EPDS) is a 10-item self-report used to measure postpartum depression with score range 0-30, a higher score indicates greater symptom burden. A score of > 6 is indicative of a woman being at risk of perinatal depression.
Time Frame: Enrollment - final study visit, approximately 24 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antidepressant Medication | Interpersonal Therapy
Number analyzed (Participants) | 39 | 39
Participants | 37 | 39

7. Secondary Outcome: Number of Women With a CGI Score Decline of One Point From Baseline
Description: The Clinical Global Impression (CGI) is a 7-point scale (range 1-7) that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with the patient. Lower scores correlate with clinical improvement.
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antidepressant Medication | Interpersonal Therapy
Number analyzed (Participants) | 39 | 39
Participants | 38 | 39

8. Secondary Outcome: Percentage of Women Experiencing Anti Depressant Medication Toxicity
Description: The percentage of women who are taking the antidepressant medication who discontinue the medication due to a grade II or higher toxicity
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Number; unit: percentage of women who discontinued
Groups:
- Women Assigned to the Antidepressant Medication Arm: All women who were randomized to the medication arm
Arm/Group | Women Assigned to the Antidepressant Medication Arm
Number analyzed (Participants) | 40
percentage of women who discontinued | 0

9. Secondary Outcome: Percentage of Women Who Adhere to the Prescribed Antidepressant Medication (ADM)
Description: Percentage of women randomized to the ADM arm with adequate adherence defined as taking >90% of pills assessed by pill count and report
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Number; unit: percentage of participants
Groups:
- All Women Assigned to the Antidepressant Medication Arm: All women who were randomized to the medication arm
Arm/Group | All Women Assigned to the Antidepressant Medication Arm
Number analyzed (Participants) | 40
percentage of participants | 14

10. Secondary Outcome: Number of Women Who Adhere to the Interpersonal Therapy Arm (IPT)
Description: Number of women randomized to the IPT arm who complete all IPT sessions
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Count of Participants; unit: Participants
Groups:
- All Women Assigned to the Therapy Arm: Women who were randomized to the interpersonal therapy arm
Arm/Group | All Women Assigned to the Therapy Arm
Number analyzed (Participants) | 40
Participants | 5

11. Secondary Outcome: Acceptability of Trial Participation for Treatment of Postpartum Depression
Description: Participants completed a satisfaction survey at the final study visit addressing issues around 4 topics: (1) satisfaction with the study; (2) satisfaction with the intervention received; (3) self-perceived improvement of mental health; and (4) preference for study intervention not received. Responses were recorded using a Likert-type rating scale with the following responses: "Strongly disagree", "disagree", "neutral", "agree", and "strongly agree". For analysis purposes responses were combined into categories as follows: Agree and Strongly Agree, Disagree and Strongly Disagree, and neutral.
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Antidepressant Medication | Interpersonal Therapy
Number analyzed (Participants) | 39 | 39
Participants
  Satisfaction with the study: Strongly Agree or Agree | 39 | 39
  Satisfaction with the intervention received: Strongly Agree or Agree | 37 | 37
  Satisfaction with the intervention received: Strongly Disagree or Disagree | 2 | 2
  Self-perceived improvement of mental health: Strongly Agree or Agree | 39 | 39
  Preference for study intervention not received: Strongly Agree or Agree | 6 | 4
  Preference for study intervention not received: Neutral | 10 | 16
  Preference for study intervention not received: Strongly Disagree or Disagree | 23 | 19

12. Secondary Outcome: Changes in the Viral Load Between Study Entry and the Last Visit
Description: The mean change in the viral load will be measured between all women enrolled between the first and last visits
Time Frame: Enrollment - final visit, approximately 24 weeks after enrollment
Measure: Mean (Standard Deviation); unit: log copies/mL
Arm/Group | Antidepressant Medication | Interpersonal Therapy
Number analyzed (Participants) | 39 | 39
log copies/mL | 0.6 (4.0) | 1.6 (3.7)

ADVERSE EVENTS:
Time Frame: From the time of signing the Informed Consent through the last follow-up visit, a total of approximately 6 months.
Arm/Group | Antidepressant Medication | Interpersonal Therapy
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 9/40 | 9/40
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antidepressant Medication (N=40) | Interpersonal Therapy (N=40)
Mild Medication Toxicity - Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 0 (0) — Nausea; Abdominal pain; Diarrhea
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 9 (9)
Mild medication toxicity - Central nervous system (Nervous system disorders) | 4 (4) | 0 (0) — Headache; Lightheadedness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT04094870/Prot_SAP_000.pdf